CLINICAL TRIAL: NCT00237913
Title: A Multicenter, Randomized, Naturalistic, Open-Label Study Between Aripiprazole and Standard of Care in the Management of Community-Treated Schizophrenic Patients (Schizophrenia Trial of Aripiprazole - STAR)
Brief Title: Schizophrenia Trial of Aripiprazole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN138-152
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Olanzapine; Quetiapine Fumarate; Risperidone

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- B1 (Active Comparator)
  Interventions: Drug: Olanzapine or Quetiapine or Risperidone

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 10 - 30 mg, Once daily, 26 weeks.
  Other Names: Abilify
  Arms: A1
Drug: Olanzapine or Quetiapine or Risperidone — Olanzapine: Tablets, Oral, 5-20 mg, Once daily, 26 weeks. OR Quetiapine: Tablets, Oral, 100-800 mg, Once daily, 26 weeks. OR Risperidone: Tablets, Oral, 2-8 mg, Once daily, 26 weeks.
  Arms: B1

SUMMARY:
Aripiprazole will show improved effectiveness over the standard of care treatment with one of three atypical antipsychotics (olanzapine, quetiapine and risperidone).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Schizophrenia symptoms not optimally controlled or antipsychotic medication not well tolerated

Exclusion Criteria:

* Diagnosis of schizoaffective disorder
* Patients treatment-resistant to antipsychotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2004-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Score on the Investigator Assessment Questionnaire at week 26

SECONDARY OUTCOMES:
Clinical Global Impression scale and patient preference of medication at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Millet, MD, Principal Investigator — Centre Hospitalier Guillaume Régnier, service de Psychiatrie adultes
Locations (33):
- Local Institution, Vienna, Austria
- Local Institution, Přerov, Czechia
- Denmark (2):
  - Local Institution, Copenhagen
  - Local Institution, Hørsholm
- Local Institution, Helsinki, Finland
- France (10):
  - Local Institution, Brumath
  - Local Institution, Dole
  - Local Institution, Hénin-Beaumont
  - Local Institution, Jonzac
  - Local Institution, Nantes Orvault
  - Local Institution, Paris
  - Local Institution, Reims
  - Local Institution, Rennes
  - Local Institution, Toulouse
  - Local Institution, Uzès
- Germany (5):
  - Local Institution, Duisburg
  - Local Institution, Hattingen
  - Local Institution, München
  - Local Institution, Nuremberg
  - Local Institution, Oldenburg
- Local Institution, Murcia, Spain
- Sweden (5):
  - Local Institution, Bromma
  - Local Institution, Gothenburgh
  - Local Institution, Halmstad
  - Local Institution, Malmo
  - Local Institution, Säter
- United Kingdom (7):
  - Local Institution, Belfast, Antrim
  - Local Institution, London, Greater London
  - Local Institution, Royal Tunbridge Wells, Kent
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Davyhulme, Lancashire
  - Local Institution, South Wales, Mid Glamorgan
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- [Derived] Hanssens L, L'Italien G, Loze JY, Marcus RN, Pans M, Kerselaers W. The effect of antipsychotic medication on sexual function and serum prolactin levels in community-treated schizophrenic patients: results from the Schizophrenia Trial of Aripiprazole (STAR) study (NCT00237913). BMC Psychiatry. 2008 Dec 22;8:95. doi: 10.1186/1471-244X-8-95. PMID 19102734